CLINICAL TRIAL: NCT07055503
Title: The αO2-PRBC.Thal Study on the Use of Hemanext One® RBC Storage System for Blood Transfusion Support on Transfusion-dependent Thalassemia
Brief Title: Use of the Hemanext One® Hypoxic Red Blood Cell Storage System for Transfusion in Thalassemia Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: University Research Institute for the Study of Genetic & Malignant Disorders in Childhood (Other)
Collaborators: Hemanext (Industry); Laikο General Hospital, Athens (Other)
Responsible Party: Principal Investigator, Antonis Kattamis, Professor of Pediatric Hematology/Oncology Head, Division of f Pediatric Hematology/Oncology First Department of Pediatrics - National & Kapodistrian University of Athens, 'Aghia Sophia' Children's Hospital, National and Kapodistrian University of Athens
Other Study IDs: αO2-PRBC.Thal
Record Dates: First submitted 2025-05-28; First posted 2025-07-09 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Transfusion-dependent Beta-Thalassemia; Blood Transfusion
Keywords: Red Blood Cell Transfusion; Anemia; Quality of Life
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Peripheral blood samples will be collected and retained for future biochemical, metabolic, and hematological analyses. Samples may be used to assess markers related to hemolysis, erythropoiesis, oxidative stress, and red blood cell metabolism. No DNA will be extracted from the retained samples. All samples will be coded and stored under secure conditions in compliance with data protection regulations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Transfusion-dependent thalassemia (TDT) requires lifelong, regular red blood cell (RBC) transfusions. Conventionally stored RBCs develop biochemical and structural "storage lesions," driven largely by oxidative stress, which may reduce post-transfusion survival and contribute to anemia, hemolysis, metabolic abnormalities, and iron overload. Hypoxic storage has emerged as a strategy to mitigate oxidative deterioration and preserve RBC quality.

The Hemanext One® system allows processing and storage of RBCs under hypoxic conditions (low oxygen and carbon dioxide). Early studies have shown improved metabolic preservation compared with standard storage. In Greece, and specifically at the National Center for Blood Transfusion (EKEA), hypoxically stored RBCs have already been introduced into routine transfusion practice for selected TDT patients, independently of this study.

This study is observational and does not assign or provide Hemanext-processed RBCs. Instead, it aims to systematically evaluate the hematologic, metabolic, and clinical impact of receiving hypoxically stored RBCs in adult TDT patients who are already being transfused with Hemanext units as part of their clinical care.

The study includes a 12-week baseline period based on conventional transfusions, followed by a treatment phase of at least 3 months during which patients continue receiving Hemanext-processed RBCs as provided by EKEA; the treatment phase may be extended for each participant up to the study-wide data cut-off date. Informed consent is obtained before any study-related data collection.

The primary objective is to compare transfusion burden (cc/kg) between baseline conventional RBCs and hypoxically stored RBCs administered in routine care. Secondary objectives include changes in pre-transfusion hemoglobin, total hemoglobin mass, hemolysis and erythropoiesis markers, metabolic indicators, iron overload parameters, quality of life, and safety outcomes. Findings will provide real-world evidence on the feasibility and clinical impact of hypoxically stored RBCs in chronically transfused patients.

DETAILED DESCRIPTION:
Transfusion-dependent β-thalassemia (TDT) is a severe inherited hemoglobinopathy requiring lifelong red blood cell (RBC) transfusions every 2 to 4 weeks. Patients typically receive 2-4 units per month, and their long-term survival and quality of life depend on the safety and functional integrity of the transfused RBCs. During standard storage, RBCs undergo progressive biochemical and morphological deterioration known as "storage lesions," which include oxidative damage, protein oxidation, enzymatic dysfunction, membrane remodeling, depletion of 2,3-diphosphoglycerate (2,3-DPG), and metabolic instability. These alterations reduce post-transfusion RBC survival and oxygen-delivery capacity and may contribute to hemolysis, increased transfusion requirements, iron accumulation, and other clinical complications. Oxygen exposure during storage is a major driver of oxidative injury, and reducing oxygen levels has been shown to mitigate the severity of storage lesions.

The Hemanext One® RBC Processing and Storage System is designed to reduce and maintain low oxygen and carbon dioxide levels during storage, thereby limiting oxidative deterioration of stored RBCs. Preclinical and early clinical evaluations have demonstrated improved preservation of RBC membrane integrity, metabolic profiles, and functional stability compared with conventional storage. The system has received FDA De Novo marketing authorization and CE marking. In Greece, RBC units processed with Hemanext One® are already used at the National Center for Blood Transfusion (EKEA) and are provided to selected thalassemia patients as part of standard clinical practice, independently of this study.

This study is prospective, observational, and entirely non-interventional. The investigators do not influence or assign transfusion type. All patients receive blood units according to routine clinical practice at EKEA, and participation in the study begins only after the patient signs informed consent. No study procedures or assessments occur before consent is obtained.

The study includes a 12-week baseline period, based on retrospective or prospectively collected routine clinical data during which the patient received conventionally stored RBCs. This is followed by an observational treatment period during which patients continue to receive hypoxically stored RBCs processed with the Hemanext One® system, exactly as provided by EKEA. The duration of this treatment observation phase is at least three months and may be extended until the study-wide data cut-off date, depending on RBC availability and patient preference. The study does not modify transfusion thresholds, clinical decision-making, or transfusion scheduling.

The primary objective of the study is to assess changes in transfusion burden, measured in cc/kg, after the transition from conventionally stored to hypoxically stored RBCs. Secondary objectives include the evaluation of changes in pre-transfusion hemoglobin, hemolysis and erythropoiesis markers, metabolic indicators, iron overload indices such as serum ferritin, patient-reported quality of life using validated instruments including the FACIT-F version 4 questionnaire, and the frequency and nature of transfusion-related adverse events. All information is obtained exclusively from routine clinical assessments and standard laboratory evaluations. No additional blood draws or study-specific procedures are required. A subset of patients may voluntarily contribute residual blood samples for more detailed laboratory evaluation, provided that these analyses are within the scope of routine laboratory capabilities.

All collected data will be coded and managed according to applicable data protection regulations. The investigators will not influence the assignment of blood unit type, which remains the responsibility of the transfusion service. This real-world evidence study aims to generate clinically meaningful insights into the safety, feasibility, and effectiveness of hypoxically stored RBCs in patients with TDT, supporting future evidence-based evaluation of their use in chronically transfused populations.

ELIGIBILITY:
Inclusion Criteria

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject is ≥ 18 years of age at the time of signing the informed consent form (ICF).
2. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
3. Subject has documented diagnosis of β- transfusion dependent thalassemia, defined as ect: ≥ 6 RBC units/24 weeks and no transfusion-free period for ≥ 42 days during the 24 weeks prior enrollment.
4. Transfusion history (including units or cc) for at least 6 months prior to enrollment needs to be available.
5. Subject is on chelation therapy and a fairly stable dose for at least 6 months prior to enrollment.
6. Chronic therapies (including hydroxyurea) are allowed as long as the medication dose has been stable for at least 6 months prior to enrollment.
7. Having been exposed to PRBC transfusions prepared with the Hemanext One processing system

Exclusion Criteria

The presence of any of the following will exclude a subject from enrollment:

1. Subject has currently or has a history of any significant medical condition, laboratory abnormality, or psychiatric illness.
2. Subject has had positive Coombs (antiglobulin) test anytime during the 6 months prior to enrollment.
3. Subject is scheduled to undergo or has recently (in the last 6 months) undergone splenectomy.
4. Use of luspatercept during the period of 6 months prior to enrollment and during the trial is not allowed.
5. Participation in an interventional clinical trial or use of experimental medications during the period of 6 months prior to enrollment and during the trial is not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults aged 18 years or older diagnosed with β-transfusion dependent thalassemia (TDT) who require regular red blood cell (RBC) transfusions, defined as receiving at least 6 units of RBCs over 24 weeks without a transfusion-free interval longer than 42 days. Participants must have a documented transfusion history and be on a stable chelation therapy regimen for at least six months prior to enrollment. Patients receiving stable doses of chronic therapies, including hydroxyurea, are eligible. Individuals with significant medical, laboratory, or psychiatric conditions that may interfere with study participation, or with a positive Coombs test within six months prior to enrollment, are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in RBC transfusion burden | Up to 6 months
  Changes from baseline in RBC transfusion burden. Significant changes are defined as a difference of >20% from baseline, corresponding to at least 1 unit per 24 weeks.

SECONDARY OUTCOMES:
Change from baseline in pre-transfusion hemoglobin. | Up to 6 months
  Assessed at each transfusion visit and compared to baseline average.
Change from baseline in fatigue-related quality of life using FACIT-F Version 4 | Week 13, Week 24
  Fatigue-related quality of life will be assessed using the FACIT-Fatigue Scale (FACIT-F v4), a validated 13-item questionnaire. Scores range from 0 to 52, with higher scores indicating less fatigue and therefore better quality of life. Changes from Week 13 and 24 will be reported as mean (±SD) score differences.
Healthcare resource utilization | Up to 6 months
  Includes number of hospital visits, admissions, and emergency care related to transfusion needs.
Change from baseline in reticulocyte count | Up to 6 months
  Reticulocyte percentage (%) will be measured at each visit and summarized as mean change from baseline.
Change from baseline in total bilirubin levels | Up to 6 months
  Total bilirubin (mg/dL) will be assessed as a marker of hemolysis. Mean changes from baseline will be summarized.
Change from baseline in lactate dehydrogenase (LDH) levels | Up to 6 months
  LDH (U/L) will be measured at regular intervals. Changes from baseline values will be reported as mean (±SD) at each visit.
Change from baseline in serum ferritin levels | Up to 6 months
  Serum ferritin (ng/mL) will be measured at defined study time points. Mean and standard deviation of changes from baseline will be reported at each visit.
Change from baseline in transferrin saturation | Up to 6 months
  Transferrin saturation (%) will be calculated from serum iron and TIBC and summarized as change from baseline.
Frequency of adverse events (AEs) | Up to 6 months
  The total number and percentage of participants experiencing one or more adverse events will be recorded. Events will be categorized by type and system organ class (SOC) according to MedDRA terminology.
Severity and seriousness of adverse events | Up to 6 months
  Severity will be graded according to CTCAE v5.0 criteria (Grade 1-5). Seriousness will be defined per ICH-GCP guidelines. Events will be reported as frequency and percentage by grade and seriousness classification.
Relationship of adverse events to Hemanext transfusion | Up to 6 months
  Each AE will be assessed for relatedness to the investigational product (Hemanext RBC unit) by the site investigator as "Not related", "Possibly related", or "Probably related". Results will be summarized descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Antonis Kattamis, Professor, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- Aghia Sophia Children's Hospital, Athens, Attica, Greece

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT07055503/Prot_SAP_002.pdf